CLINICAL TRIAL: NCT01753414
Title: POSTILV: A RANDOMIZED PHASE II TRIAL IN PATIENTS WITH OPERABLE STAGE I NON-SMALL CELL LUNG CANCER: RADICAL RESECTION VERSUS ABLATIVE STEREOTACTIC RADIOTHERAPY - This is a Limited Participation Study.
Brief Title: Radical Resection Vs. Ablative Stereotactic Radiotherapy in Patients With Operable Stage I NSCLC
Acronym: POSTILV
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RF-3502
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Radiosurgery; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery (Other): R0 resection (radical resection) with nodal dissection or sampling (RODS).
  Interventions: Procedure: Surgery
- Stereotactic Body Radiation Therapy (SBRT) (Experimental): Stereotactic Body Radiation Therapy (SBRT) given every other day 11 Gy in 5 fractions to a total dose of 55 Gy in 10-15 days with an inter-fraction interval of 2-3 days.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Daily fractions
  Arms: Stereotactic Body Radiation Therapy (SBRT)
Procedure: Surgery — Radical resection
  Arms: Surgery

SUMMARY:
Rationale: Surgery remains the standard of care for stage 1 (T1-2a N0)non-small cell lung cancer. Stereotactic body radiation therapy is a newer radiation treatment that gives fewer but higher and possibly more effective doses of radiation than standard radiation. This technique may be able to send x-rays directly to the tumor and cause less damage to normal tissue. It is not yet known whether stereotactic body radiation therapy is more effective than surgery in treating non-small cell lung cancer.

Purpose: The primary aim of this randomized phase II trial is to determine if the efficacy of SBRT is comparable to that of standard surgical interventions for patients with T1N0 non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

- Pathologically (histologically or cytologically) proven diagnosis of Stage I NSCLC [American Joint Committee on Cancer (AJCC), 7th ed.], T1N0M0; note: T1N0 disease must be confirmed by FDG-PET/CT. (FDG = 18F-fluorodeoxyglucose; PET = positron emission tomography; CT = Computed Tomography)

Biopsy confirmation of diagnosis is strongly recommended but not required. If the biopsy is attempted and non-diagnostic, if the patient refuses biopsy, or if the risk of biopsy is considered too high, patients may be enrolled if the mass is suspicious for NSCLC based on 2 or more of the following criteria:

* Positive smoking history;
* Absence of benign calcifications within suspicious nodule;
* Activity on PET greater than normal tissue;
* Evidence of growth compared to previous imaging;
* Presence of spiculation.

The following primary cancer types are eligible: squamous cell carcinoma; adenocarcinoma; large cell carcinoma/ large cell neuroendocrine carcinoma; non-small cell carcinoma not otherwise specified.

* Patients with hilar or mediastinal lymph nodes ≤ 1 cm and no abnormal hilar or mediastinal uptake on PET and CT will be considered N0. Mediastinal lymph node biopsy is required for patients with visible nodes: patients with > 1 cm hilar or mediastinal lymph nodes on CT or with nodes appearing as abnormal on PET (including suspicious but nondiagnostic uptake). Such patients will not be eligible unless directed biopsies of all abnormal lymph nodes are negative for cancer or these nodes demonstrate a lack of change during the prior 6 months and thus are considered to be non-malignant.
* The patient must be considered a reasonable candidate for surgical resection using a lobectomy or pneumonectomy of the primary tumor within 6 weeks prior to registration, according to the following criteria based on the American College of Chest Physicians guidelines [165]:

  * A qualified thoracic surgeon should make the determination that there would be a high likelihood of negative surgical margins;
  * Baseline forced expiratory volume in 1 second (FEV1) >60% predicted, postoperative predicted FEV1 >40% predicted;
  * Diffusion capacity of the lung for carbon monoxide (DLCO) >60% predicted, postoperative predicted DLCO > 40 % predicted;
  * No baseline hypoxemia and/or hypercapnia;
  * If the estimated postoperative FEV1 or DLCO <40% predicted indicates an increased risk for perioperative complications, including death, from a standard lung cancer resection (lobectomy or greater removal of lung tissue), then cardiopulmonary exercise testing to measure maximal oxygen consumption (VO2max) must be >60%;
  * No severe pulmonary hypertension;
  * No severe cerebral, acute or chronic cardiac, or peripheral vascular disease;
* Pleural effusion, if present, must be deemed too small to tap under CT guidance and must not be evident on chest x-ray. Pleural effusion that appears on chest x-ray will be permitted only if there is no evidence of malignancy after invasive cytologic assessment.
* Appropriate stage for protocol entry, including no distant metastases, based upon the following minimum diagnostic workup:

  * History/physical examination, including documentation of weight within 6 weeks prior to registration;
  * Evaluation by an experienced thoracic surgeon within 6 weeks prior to registration;
  * FDG-PET/CT scan for staging and RT plan within 4 weeks prior to registration;
  * CT scan (preferably with intravenous contrast, unless medically contraindicated) within 4 weeks prior to registration to include the entirety of both lungs, the mediastinum, liver, and adrenal glands; primary tumor dimension will be measured on CT scan.
* Zubrod Performance Status 0-1 within 6 weeks prior to registration;
* Age ≥ 18;
* For women of childbearing potential, a serum or urine pregnancy test must be negative within 72 hours prior to registration;
* Women of childbearing potential and male participants who are sexually active must practice adequate contraception during treatment if assigned to treatment with SBRT.
* Patients must provide study specific informed consent prior to study entry.

Exclusion Criteria:

* Direct evidence of regional or distant metastases after PET and surgical staging studies, or synchronous primary malignancy or prior invasive malignancy in the past 3 years, with the following exceptions:

  * carcinoma in situ;
  * early stage skin cancer that has been definitively treated;
  * when an invasive malignancy has been treated definitively and the patient has remained disease free for ≥ 3 years;
* Primary tumors >3 cm;
* Prior systemic chemotherapy or thoracic surgery involving lobectomy or pneumonectomy;
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields;
* Pure bronchioloalveolar carcinoma subtype of non-small cell lung cancer;
* Active systemic, pulmonary, or pleural pericardial infection;
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-12; Primary Completion 2023-04-03 (Actual); Study Completion 2026-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Ming (Spring) Kong, MD, PhD, Principal Investigator — Case Western Reserve University
Locations (4):
- China (4):
  - Chinese Academy of Medical Science, Beijing
  - Shandong Cancer Hospital, Jinan, Shangdong
  - Shanghai Cancer Center/Fudan University, Shanghai
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Elbanna M, Shiue K, Edwards D, Cerra-Franco A, Agrawal N, Hinton J, Mereniuk T, Huang C, Ryan JL, Smith J, Aaron VD, Burney H, Zang Y, Holmes J, Langer M, Zellars R, Lautenschlaeger T. Impact of Lung Parenchymal-Only Failure on Overall Survival in Early-Stage Lung Cancer Patients Treated With Stereotactic Ablative Radiotherapy. Clin Lung Cancer. 2021 May;22(3):e342-e359. doi: 10.1016/j.cllc.2020.05.024. Epub 2020 Jun 2. PMID 32736936

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 47 participants registered to the first step of the study, 44 were randomized. Randomization required FDG-PET/CT (FDG = 18F-fluorodeoxyglucose; PET = positron emission tomography; CT = Computed Tomography) staging to confirm T1N0 disease, per American Joint Committee on Cancer (AJCC), 7th edition.
Period: Overall Study
Arm/Group | Surgery | Stereotactic Body Radiation Therapy (SBRT)
Started | 22 | 22
Completed (Participants contributing data to results are considered to have completed the study.) | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgery | Stereotactic Body Radiation Therapy (SBRT) | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Median (Full Range); unit: years] | 62.5 [49 to 78] | 67 [59 to 82] | 65 [49 to 82]
Age, Customized [Count of Participants; unit: Participants]
  <50 | 1 | 0 | 1
  50-59 | 6 | 1 | 7
  60-69 | 11 | 13 | 24
  70-79 | 4 | 6 | 10
  ≥80 | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 13 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 22 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 22 | 22 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 22 | 22 | 44
Zubrod performance status [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound; 5 = Death
  Participants
    0 | 6 | 5 | 11
    1 | 16 | 17 | 33
Histology [Count of Participants; unit: Participants]
  Squamous cell carcinoma | 4 | 5 | 9
  Adenocarcinoma | 14 | 12 | 26
  Non-small cell caarcinoma, NOS | 4 | 5 | 9
Forced expiratory volume in one second (FEV1) [Median (Full Range); unit: liters/second] | 2.31 [1.6 to 3.82] | 2.15 [1.3 to 3.33] | 2.29 [1.3 to 3.82]
Percent predicted FEV1 [Median (Full Range); unit: percentage] — Percentage of the predicted normal value based on age, gender, height, and ethnicity. Higher value indicates better condition. Population: Randomized participants with data
  percentage
    number analyzed (Participants) | 22 | 21 | 43
    (all) | 96.1 [62 to 133] | 90 [62 to 129.2] | 94 [62 to 133]
Forced vital capacity (FVC) [Median (Full Range); unit: liters/second] | 3.2 [2.2 to 4.79] | 2.855 [1.59 to 4.42] | 2.96 [1.59 to 4.79]
Percent predicted FVC [Median (Full Range); unit: percentage] — Percentage of the predicted normal value based on age, gender, height, and ethnicity. Higher value indicates better condition. Population: Randomized participants with data
  percentage
    number analyzed (Participants) | 22 | 21 | 43
    (all) | 99 [65 to 133] | 98.7 [66.5 to 140.1] | 98.7 [65 to 140.1]
Percent predicted Diffusing capacity for carbon monoxide (DLCO) [Median (Full Range); unit: percentage] — Percentage of the predicted normal value based on age, gender, height, and ethnicity. Higher value indicates better condition. Population: Randomized participants with data
  percentage
    number analyzed (Participants) | 22 | 20 | 42
    (all) | 90 [62 to 190] | 89 [65 to 102] | 90 [62 to 190]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Alive Without Local-regional Failure at Two Years (Local-regional Tumor Control)
Description: Local-regional failure (LRF) is defined differently for each arm. LRF after RODS is defined as recurrence, defined by CT, confirmed by PET/CT whenever possible, i.e., development of tumor masses at site of resection, hilum (N1 nodal region), mediastinum (N2-N3 nodes), ipsilateral supraclavicular fossa for upper lobe tumors (N3 nodes), or within 3 cm of the staple line of RODS. LRF after SBRT is defined as tumor progression on CT per Response Evaluation Criteria in Solid Tumors (RECIST) criteria, confirmed by positron PET/CT, within same lobe, hilum (N1 nodes), mediastinum (N2-N3 nodes), or ipsilateral supraclavicular fossa for upper lobe tumors (N3 nodes), or within 3 cm of original planning target volume (PTV). Local-regional control time is defined as time from randomization to the date of first LRF, death, or last known follow-up (censored), whichever occurred first. Rates are estimated using the Kaplan-Meier method.
Time Frame: From date of randomization to two years
Population: Randomized participants with follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 21 | 21
percentage of participants | 95.2 [70.7 to 99.3] | 66.7 [42.5 to 82.5]

2. Secondary Outcome: Overall Survival (Percentage of Participants Alive)
Description: Overall survival rates are estimated by the Kaplan-Meier method. The distribution of DFS estimates between the two arms is compared using the log rank test. Overall survival time is defined as time from randomization to the date of death from any cause or last known follow-up (censored). Two-year rates are provided.
Time Frame: From date of randomization to date of death or last follow-up. Maximum follow-up was 7.0 years.
Population: Randomized participants with follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 21 | 21
percentage of participants | 85.7 [62.0 to 95.2] | 90.5 [67.0 to 97.5]

3. Secondary Outcome: Percentage of Participants With Local-regional Failure (LRF)
Description: LRF rates are estimated using the cumulative incidence method. LRF is defined differently for each arm. LRF after RODS is defined as recurrence, defined by CT, confirmed by PET/CT whenever possible, i.e., development of tumor masses at site of resection, hilum (N1 nodal region), mediastinum (N2-N3 nodes), ipsilateral supraclavicular fossa for upper lobe tumors (N3 nodes), or within 3 cm of the staple line of RODS. LRF after SBRT is defined as tumor progression on CT per Response Evaluation Criteria in Solid Tumors (RECIST) criteria, confirmed by PET/CT, within same lobe, hilum (N1 nodes), mediastinum (N2-N3 nodes), or ipsilateral supraclavicular fossa for upper lobe tumors (N3 nodes), or within 3 cm of original PTV. LRF time is defined as time from randomization to the date of first LRF, last known follow-up (censored), or death without LRF (competing risk), whichever occurred first. Two-year rates are provided.
Time Frame: From date of randomization to the date of first local-regional failure, death, or last known follow-up, whichever occurred first. Maximum follow-up is 7.0 years.
Population: Randomized participants with follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 21 | 21
percentage of participants | 4.8 [0.3 to 20.2] | 33.3 [14.4 to 53.6]

4. Secondary Outcome: Percentage of Participants With Distant Failure
Description: Distant failure rates are estimated using the cumulative incidence method. Distant failure is defined as appearance of tumor within another ipsilateral (non-primary) lobe ≥ 2 cm from the original planning target volume (PTV) or distant metastasis, including appearance of tumor deposits characteristic of NSCLC metastasis (chest wall other than incision sites, mediastinal structures/diaphragm, malignant pleural/pericardial effusion), contralateral lung and/or other distant sites. Time to distant failure is defined as time from randomization to the date of first failure, last known follow-up (censored), or death without failure (competing risk). Two-year rates are provided.
Time Frame: From date of randomization to date of first distant failure, death, or last known follow-up, whichever occurred first. Maximum follow-up was 7.0 years.
Population: Randomized participants with follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 21 | 21
percentage of participants | 23.8 [8.3 to 43.6] | 23.8 [8.4 to 43.6]

5. Secondary Outcome: Percentage of Participants Alive Without Disease [Disease-free Survival (DFS)]
Description: Failure rates are estimated using the Kaplan-Meier method, where failure is defined as LRF, DF, or death from any cause. LRF is defined differently for each arm. LRF after RODS is defined as recurrence, defined by CT, confirmed by PET/CT whenever possible, i.e., development of tumor masses at the resection site, hilum, mediastinum, or ipsilateral supraclavicular fossa for upper lobe tumors, or within 3 cm of the staple line of RODS. LRF after SBRT is defined as tumor progression on CT per RECIST criteria, confirmed by PET/CT, within same lobe, hilum, mediastinum, or ipsilateral supraclavicular fossa for upper lobe tumors, or within 3 cm of original PTV. DF is defined as tumor within a non-primary lobe ≥ 2 cm from the original planning target volume or distant metastasis. Failure time is defined as time from randomization to the date of first failure or last known follow-up (censored), whichever occurred first. Two-year rates are provided.
Time Frame: From date of randomization to the date of first failure, death, or last known follow-up, whichever occurred first. Maximum follow-up is 7.0 years.
Population: Randomized participants with follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 21 | 21
percentage of participants | 65.0 [40.3 to 81.5] | 61.9 [38.1 to 78.8]

6. Secondary Outcome: Number of Participants by Failure Site
Description: Local-regional failure (LRF) is defined differently for each arm. LRF after RODS is defined as recurrence, defined by CT, confirmed by PET/CT whenever possible, i.e., development of tumor masses at site of resection, hilum, mediastinum, ipsilateral supraclavicular fossa for upper lobe tumors, or within 3 cm of the staple line of RODS. LRF after SBRT is defined as tumor progression on CT per RECIST criteria, confirmed by PET/CT, within same lobe, hilum, mediastinum, or ipsilateral supraclavicular fossa for upper lobe tumors, or within 3 cm of original planning target volume (PTV). Distant failure is defined as tumor within a non-primary lobe ≥ 2 cm from the original planning target volume or distant metastasis, including tumor deposits characteristic NSCLC metastasis (chest wall other than incision sites, mediastinal structures/diaphragm, malignant pleural/pericardial effusion), contralateral lung and/or other distant sites.
Time Frame: From date of randomization to date of last known follow-up. Maximum follow-up was 7.0 years.
Population: Randomized participants with follow-up data
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 21 | 21
Participants
  Local-regional failure (at any time) | 2 | 9
  Distant failure (at any time) | 6 | 7

7. Secondary Outcome: Best PET Tumor Response
Description: PET Tumor Response of Irradiated Target Lesions is defined as
  * Complete Metabolic Response (CMR): Tumor 18F-fluorodeoxyglucose (FDG)-activity decreased to less than mean background of the aortic arch blood pool.
  * Partial Metabolic Response (PMR): At least a 30% decrease in the maximum of relative tumor FDG-activity of target lesions
  * Progressive Metabolic Disease (PMD): At least a 20% increase in the maximum of relative tumor FDG-activity of target lesions
  * Stable Metabolic Disease (SMD): Neither sufficient reduction to qualify for (major pathological response) PMR nor sufficient increase to qualify for PMD The percentage of decrease or increase was globally estimated based on readings of (tumor activity-aorta activity)/aorta activity.
Time Frame: From date of randomization to date of last known follow-up. Maximum follow-up was 7.0 years.
Population: Randomized participants with follow-up PET scan
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 3 | 4
Participants
  Complete Metabolic Response | 0 | 0
  Partial Metabolic Response | 0 | 0
  Progressive Metabolic Disease | 3 | 4
  Stable Metabolic Disease | 0 | 0

8. Secondary Outcome: Number of Participants by Highest Grade Adverse Event Reported
Description: Common Terminology Criteria for Adverse Events (version 4.0) grades adverse event severity from 1=mild to 5=death. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: From date of randomization to the date of last known follow-up. Maximum follow-up time was 7.0 years.
Population: Randomized participants who started protocol treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 16 | 19
Participants
  Grade 1 | 7 | 11
  Grade 2 | 6 | 3
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

9. Secondary Outcome: Number of Participants With Surgical and Radiation Treatment Credentialing Completed and Documented Before Enrollment (Trial Feasibility)
Time Frame: baseline
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 22 | 22
Participants | 22 | 22

10. Secondary Outcome: Number of Eligible Participants (Trial Feasibility)
Description: Goal: 95% of participants retain eligibility status (meet all eligibility criteria) after central review by headquarters staff.
Time Frame: Baseline
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 22 | 22
Participants | 17 | 14

11. Secondary Outcome: Number of Participants With Baseline Forms Completed and Provided Within 30 Days of Randomization (Trial Feasibility)
Time Frame: Baseline
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 22 | 22
Participants | 12 | 6

12. Secondary Outcome: Number of Participants Lost to Follow-up (Trial Feasibility)
Description: Goal: < 3% of participants lost to follow-up.
Time Frame: From date of randomization to date of last known follow-up. Maximum follow-up was 7.0 years.
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 22 | 22
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Baseline to the date of last known follow-up. Maximum follow-up time was 7.0 years.
Description: All-cause mortality was assessed in randomized participants with follow-up data. Adverse events were assessed in randomized participants who started protocol treatment.
Arm/Group | Surgery | Stereotactic Body Radiation Therapy (SBRT)
All-Cause Mortality (participants affected / at risk) | 5/21 | 5/21
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/19
Other Adverse Events (participants affected / at risk) | 13/16 | 15/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Surgery (N=16) | Stereotactic Body Radiation Therapy (SBRT) (N=19)
Anemia (Blood and lymphatic system disorders) | 7 | 3
Constipation (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Fever (General disorders) | 0 | 1
Pain (General disorders) | 7 | 1
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 10 | 0
Activated partial thromboplastin time prolonged (Investigations) | 4 | 2
Alanine aminotransferase increased (Investigations) | 4 | 2
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 1
Blood bilirubin increased (Investigations) | 3 | 7
CPK increased (Investigations) | 2 | 0
Cardiac troponin T increased (Investigations) | 1 | 0
Cholesterol high (Investigations) | 4 | 4
Lymphocyte count decreased (Investigations) | 1 | 5
Platelet count decreased (Investigations) | 2 | 2
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 0 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 3 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 2 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Hemoglobinuria (Renal and urinary disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 13 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 10 | 15

LIMITATIONS AND CAVEATS:
This study stopped accrual early due to unmet targeted accrual goals with 44 participants randomized out of 72 planned. Statistical testing was not done due to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT01753414/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT01753414/ICF_001.pdf